CLINICAL TRIAL: NCT03858101
Title: An Exploratory Matched Case-control Study to Measure Blood Nutrient Levels of Adult PKU Patients on a Protein Substitute.
Brief Title: SNAP: Study Nutrients in Adult PKU
Acronym: SNAP
Status: Completed | Type: Observational
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: MBB16TA10778
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2021-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PKU subjects
- Age and sex-matched non-PKU comparison subjects

SUMMARY:
Phenylketonuria (PKU) is a rare inherited metabolic disorder, where subjects are born with a genetic deficiency in the phenylalanine hydroxylase enzyme (PAH), which leaves them unable to convert Phenylalanine (Phe) into Tyrosine (Tyr). PKU patients have specific dietary needs and must follow a restrictive diet in the aim of preventing toxic levels of the amino acid phenylalanine (Phe) accumulation.

DETAILED DESCRIPTION:
The aim of this explorative cross-sectional study is to gain quantitative insights on blood nutrient levels of adult PKU patients on a protein substitute.

ELIGIBILITY:
- Inclusion Criteria:

Both PKU and Non-PKU comparison subjects:

1. Age ≥18 years
2. Willing and able to provide signed informed consent PKU specific inclusion criteria
3. PKU patients identified by newborn screening and started low Phe diet before 1 month age
4. Usage of at least one Phe-free protein substitute (i.e. an amino acid mixture including micronutrients) on a daily basis for at least 26 consecutive weeks up to Visit 1

   Non-PKU comparison subjects specific inclusion criteria:
5. Same age- (±3 years) and sex as an included PKU subject

   * Exclusion Criteria:

Both PKU and Non-PKU comparison subjects:

1. For women: Currently pregnant or lactating
2. Current psychiatric disorders
3. Current Substance Use Disorders (as described in DSM V)
4. Current use of psychotropic and/or inotropic medication
5. Omega-3, antioxidant, (multi)vitamin and/or (multi)mineral supplement use within six weeks prior to entry in the study
6. Severe hepatic, thyroid or renal dysfunction
7. No acute illnesses like flu, diarrhea, or vomiting (subjects should be symptom free for a week prior to V1)
8. Participation in any other clinical intervention studies involving test products concomitantly or within six weeks prior to entry into the study
9. Other family members taking part in this study

   PKU subject specific exclusion criteria:
10. Use of BH4, or drugs that may interfere with main outcomes

    Non-PKU comparison subjects specific exclusion criteria:
11. Any condition or special diet (e.g. vegan or vegetarian diet) that effects the metabolism and/or normal dietary pattern/intake
12. A first or second degree relative with inborn errors of metabolism
13. Living together with someone with inborn errors of metabolism (e.g. partner, spouse or roommate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PKU subjects (18 years and olders) and non PKU comparisons.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Blood nutritional status | day 1
  Micro-and macronutrients and amino acid levels [in a.o. mg/L]

SECONDARY OUTCOMES:
Blood nutritional status | day 1
  Phe/Tyr ratio [µmol/L]
Nutrient intake | day 1 - day 7
  measured by three-day food diary. Nutrients in [mg/day]
Subjective cognitive well-being | day 1 - day 7
  measured by FACT-Cog questionnaire: [four domains [score-range): 1) patients' perceived cognitive impairments [0-80]; 2) perceived cognitive abilities [0-36]; 3) noticeability or comments from others [0-16]; 4) impact of cognitive changes on quality of life [0-16]. A summary score is obtained by summing all item scores [0-148].

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Gent, Ghent, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Spain (2):
  - Úniversity Clinical Hospital, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No